CLINICAL TRIAL: NCT00061594
Title: A Phase III, Multicenter, Randomized, Double Masked, Active Treatment-Controlled Study of the Efficacy and Safety of rhuFab V2 (Ranibizumab) Compared With Verteporfin (Visudyne) Photodynamic Therapy in Subjects With Predominantly Classic Subfoveal Neovascular Age-Related Macular Degeneration
Brief Title: A Study to Compare rhuFab V2 With Verteporfin Photodynamic in Treating Subfoveal Neovascular Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FVF2587g
Record Dates: First submitted 2003-05-29; First posted 2003-05-30 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Macular Degeneration
Keywords: Neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

INTERVENTIONS:
Drug: rhuFab V2 (ranibizumab)

SUMMARY:
This is a phase III, multicenter, randomized, double-masked, active treatment-controlled study of intravitreally administered ranibizumab compared with verteporfin (Visudyne) photodynamic therapy (PDT) in treating subfoveal neovascular mascular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >=50 years
* Eligibility for treatment with PDT using verteporfin in the study eye according to the Visudyne product labeling
* Future treatment with PDT using verteporfin anticipated or expected in the study eye
* Primary or recurrent subfoveal choroidal neovascularization (CNV) lesions secondary to age-related macular degeneration (AMD) in the study eye
* A classic CNV component (well-demarcated hyperfluorescence boundaries in the early phase of the fluorescein angiogram) that is >=50% of the total lesion size
* Total lesion size of less than or equal to 5400 um in greatest linear dimension (GLD)
* Best corrected visual acuity, using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts, of 20/40 to 20/320 (Snellen equivalent) in the study eye

Exclusion Criteria:

* Prior treatment with verteporfin, external-beam radiation therapy, or transpupillary thermotherapy (TTT) in the study eye
* Treatment with verteporfin in the non-study eye less than 7 days preceding Day 0
* Previous participation in a clinical trial (for either eye) involving anti angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)
* Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Day 0
* History of vitrectomy surgery in the study eye
* History of submacular surgery or other surgical intervention for AMD in the study eye
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)
* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either >=50% of the total lesion area or >=1 disc area (DA) in size
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the Investigator could either: (1) Require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition, or (2) If allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 24-month study period
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >=30 mmHg despite treatment with anti-glaucoma medication)
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Premenopausal women not using adequate contraception
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded by the central reading center
* Inability to comply with study or follow up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426
Dates: Start 2003-05; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (82):
- United States (70):
  - Retina Centers, P.C., Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - UC Irvine, Irvine, California
  - Doheny Eye Institute, Los Angeles, California
  - California Vitreoretinal Research Center, Menlo Park, California
  - No. California Retina-Vitreous Associates, Mountain View, California
  - UCSF School of Medicine, San Francisco, California
  - Danbury Eye Physicians & Surgeons, Danbury, Connecticut
  - New England Retina Associates, Hamden, Connecticut
  - Florida Retina Institute, Daytona Beach, Florida
  - Retina Vitreous Consultants, Fort Lauderdale, Florida
  - Retina Consultants of Southwest Florida, Fort Myers, Florida
  - Retina Health Center, Fort Myers, Florida
  - Retina Associates of South Florida, Margate, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Central Florida Retina, Orlando, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Ophthalmic Consultants, Sarasota, Florida
  - Southern Vitreoretinal Associates PA, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Thomas A. Ciulla, MD, PC, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Retina Associates PC, Annapolis, Maryland
  - New England Eye Center, Boston, Massachusetts
  - Center for Eye Research, Boston, Massachusetts
  - New England Retina Consultants, West Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Associated Retinal Consultants, Grand Rapids, Michigan
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Retina Consultants of Michigan, Southfield, Michigan
  - Retina Associates of St. Louis, Florissant, Missouri
  - St. Louis University Eye Institute, St Louis, Missouri
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - Lions Eye Institute, Albany, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Western Carolina Retinal Associates, PA, Asheville, North Carolina
  - Southeast Clinical Research, Charlotte, North Carolina
  - Duke Univ Medical Center/Duke Eye Center, Durham, North Carolina
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Flavio Company, Cincinnati, Ohio
  - Cleveland Clinic Foundation/Cole Eye Institute, Cleveland, Ohio
  - Midwest Retina, Columbus, Ohio
  - Retina Vitreous Associates, Toledo, Ohio
  - Retinal Associates of Oklahoma, Oklahoma City, Oklahoma
  - Retina & Vitreous Center of So. Oregon, Ashland, Oregon
  - Pennsylvania Retina Specialists, Camp Hill, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Retina Consultants of Charleston, Charleston, South Carolina
  - Palmetto Retina Center, Columbia, South Carolina
  - BH Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Retina Vitreous Associates, Nashville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Brian Berger, MD P.A., Austin, Texas
  - Retina Specialists, DeSoto, Texas
  - UTMB, Galveston, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - Univ of Texas Health Science Center, San Antonio, Texas
  - Medical Center Ophthalmology, San Antonio, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - John Moran Eye Center/Univ of Utah, Salt Lake City, Utah
  - Retina Group of Washington, Fairfax, Virginia
  - Vitreoretinal Associates, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - University of Melbourne, Department of Ophthalmology, East Melbourne
  - Marsden Eye Research Pty Ltd, Parramatta
  - Save Sight Institute, Sydney
  - Westmead Hospital, Westmead
- Onci klinika FNKV, Prague, Czechia
- France (3):
  - Clinique d'Ophtalmologie, Créteil
  - Clinique Monticelli, Marseille
  - HÃ´pital LariboisiÃ¨re, Paris
- Germany (3):
  - UniversitÃ¤tsklinikum Bonn, Bonn
  - Universitatskliniken Koln, Cologne
  - UniversitÃ¤tsklinikum Leipzig, Leipzig
- Semmelweis University, 1st Ophthalmological Department, Budapest, Hungary

REFERENCES:
- [Result] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Result] Kaiser PK, Brown DM, Zhang K, Hudson HL, Holz FG, Shapiro H, Schneider S, Acharya NR. Ranibizumab for predominantly classic neovascular age-related macular degeneration: subgroup analysis of first-year ANCHOR results. Am J Ophthalmol. 2007 Dec;144(6):850-857. doi: 10.1016/j.ajo.2007.08.012. Epub 2007 Oct 22. PMID 17949673
- [Result] Brown DM, Michels M, Kaiser PK, Heier JS, Sy JP, Ianchulev T; ANCHOR Study Group. Ranibizumab versus verteporfin photodynamic therapy for neovascular age-related macular degeneration: Two-year results of the ANCHOR study. Ophthalmology. 2009 Jan;116(1):57-65.e5. doi: 10.1016/j.ophtha.2008.10.018. PMID 19118696
- [Result] Suner IJ, Kokame GT, Yu E, Ward J, Dolan C, Bressler NM. Responsiveness of NEI VFQ-25 to changes in visual acuity in neovascular AMD: validation studies from two phase 3 clinical trials. Invest Ophthalmol Vis Sci. 2009 Aug;50(8):3629-35. doi: 10.1167/iovs.08-3225. Epub 2009 Feb 28. PMID 19255158
- [Result] Bressler NM, Chang TS, Fine JT, Dolan CM, Ward J; Anti-VEGF Antibody for the Treatment of Predominantly Classic Choroidal Neovascularization in Age-Related Macular Degeneration (ANCHOR) Research Group. Improved vision-related function after ranibizumab vs photodynamic therapy: a randomized clinical trial. Arch Ophthalmol. 2009 Jan;127(1):13-21. doi: 10.1001/archophthalmol.2008.562. PMID 19139332
- [Derived] Thach AB, Yau L, Hoang C, Tuomi L. Time to clinically significant visual acuity gains after ranibizumab treatment for retinal vein occlusion: BRAVO and CRUISE trials. Ophthalmology. 2014 May;121(5):1059-66. doi: 10.1016/j.ophtha.2013.11.022. Epub 2014 Jan 11. PMID 24424249
- [Derived] Weinberg DV, Shapiro H, Ehrlich JS. Ranibizumab treatment outcomes in phakic versus pseudophakic eyes: an individual patient data analysis of 2 phase 3 trials. Ophthalmology. 2013 Jun;120(6):1278-82. doi: 10.1016/j.ophtha.2012.11.042. Epub 2013 Feb 28. PMID 23453513
- [Derived] Bressler NM, Chang TS, Varma R, Suner I, Lee P, Dolan CM, Ward J, Ianchulev T, Fine J. Driving ability reported by neovascular age-related macular degeneration patients after treatment with ranibizumab. Ophthalmology. 2013 Jan;120(1):160-8. doi: 10.1016/j.ophtha.2012.07.027. Epub 2012 Sep 23. PMID 23009891
- [Derived] Rosenfeld PJ, Shapiro H, Ehrlich JS, Wong P; MARINA and ANCHOR Study Groups. Cataract surgery in ranibizumab-treated patients with neovascular age-related macular degeneration from the phase 3 ANCHOR and MARINA trials. Am J Ophthalmol. 2011 Nov;152(5):793-8. doi: 10.1016/j.ajo.2011.04.025. Epub 2011 Jul 26. PMID 21794843
- [Derived] Rosenfeld PJ, Shapiro H, Tuomi L, Webster M, Elledge J, Blodi B; MARINA and ANCHOR Study Groups. Characteristics of patients losing vision after 2 years of monthly dosing in the phase III ranibizumab clinical trials. Ophthalmology. 2011 Mar;118(3):523-30. doi: 10.1016/j.ophtha.2010.07.011. PMID 20920825
- [Derived] Barbazetto IA, Saroj N, Shapiro H, Wong P, Ho AC, Freund KB. Incidence of new choroidal neovascularization in fellow eyes of patients treated in the MARINA and ANCHOR trials. Am J Ophthalmol. 2010 Jun;149(6):939-946.e1. doi: 10.1016/j.ajo.2010.01.007. Epub 2010 Apr 8. PMID 20378094
- [Derived] Bressler NM, Chang TS, Suner IJ, Fine JT, Dolan CM, Ward J, Ianchulev T; MARINA and ANCHOR Research Groups. Vision-related function after ranibizumab treatment by better- or worse-seeing eye: clinical trial results from MARINA and ANCHOR. Ophthalmology. 2010 Apr;117(4):747-56.e4. doi: 10.1016/j.ophtha.2009.09.002. Epub 2010 Mar 2. PMID 20189654